CLINICAL TRIAL: NCT01291563
Title: A Double-blind, Randomized, Placebo- and Active-controlled, Parallel-group Trial to Evaluate the Effect of Single-dose TMC207 on the QT/QTc Interval in Healthy Subjects
Brief Title: TMC207TBC1003 - A Study in Healthy Volunteers Investigating the Effect of Single-dose TMC207 on the QT/QTc Interval Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017167; TMC-207-TBC1003
Record Dates: First submitted 2011-02-01; First posted 2011-02-08 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteer
Keywords: TMC207TBC1003; TMC207; M.Tuberculosis; TBC; Moxifloxacin; ECG; QT/QTc; Healthy volunteers
MeSH Terms: interventions — Moxifloxacin; bedaquiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 001 (Experimental): TMC207 8 tablets of TMC207 (100 mg/tablet) on Day 1
  Interventions: Drug: TMC207
- 002 (Placebo Comparator): TMC207 placebo 8 tablets of TMC207 placebo on Day 1
  Interventions: Drug: TMC207 placebo
- 003 (Active Comparator): Moxifloxacin 1 capsule of moxifloxacin (400 mg/capsule) on Day 2
  Interventions: Drug: Moxifloxacin
- 004 (Placebo Comparator): Moxifloxacin placebo 1 capsule of moxifloxacin placebo on Day 2
  Interventions: Drug: Moxifloxacin placebo

INTERVENTIONS:
Drug: Moxifloxacin — 1 capsule of moxifloxacin (400 mg/capsule) on Day 2
  Arms: 003
Drug: TMC207 — 8 tablets of TMC207 (100 mg/tablet) on Day 1
  Arms: 001
Drug: TMC207 placebo — 8 tablets of TMC207 placebo on Day 1
  Arms: 002
Drug: Moxifloxacin placebo — 1 capsule of moxifloxacin placebo on Day 2
  Arms: 004

SUMMARY:
The purpose of this study is to evaluate the effect of an 800-mg single dose of TMC207 on the QT/QTc interval in healthy volunteers.

DETAILED DESCRIPTION:
TMC207 is being investigated for the treatment of M. Tuberculosis (MTB, formerly known as TBC) infection. This study is designed to establish the effect of a single dose of TMC207 on the QT/QTc interval in healthy volunteers under fed conditions. This is a Phase I, double-blind (study doctor nor participants will know which treatment will be received), randomized (study medication is assigned by chance, like tossing a coin), placebo- and active-controlled study to evaluate the effect of single-dose TMC207 on the QT/QTc interval in healthy volunteers. A single dose of 400 mg moxifloxacin will be used as a positive control to assess trial sensitivity. The trial population will consist of 88 healthy volunteers. Forty-four participants will be randomized to Group 1, and 22 participants will be randomized to each of the Groups 2 and 3. Each gender should be represented by at least 40%. Each participant will receive one of the Treatments A or B in one treatment session. Participants in Group 1 will take a single 800-mg dose of TMC207 on Day 1 and a single dose of moxifloxacin placebo on Day 2 (Treatment A). Participants in Groups 2 and 3 will take a single dose of TMC207 placebo on Day 1 and a single 400-mg dose of moxifloxacin on Day 2 (Treatment B). All intakes of TMC207, moxifloxacin, TMC207 placebo and moxifloxacin placebo will be taken with standardized meals. The duration of the study will be 3 days, screening and follow-up period not included. On Days -1, 1, and 2 of Treatment A and B, electrocardiograms (ECGs) will be recorded continuously for 24 hours per day by Holter monitoring. Safety assessments (blood and urine tests, blood pressure, pulse, electrocardiogram, and physical examination) will follow a similar schedule and will be performed during each treatment period, up to 4 weeks after the last study drug intake.The pharmacokinetic characteristics (level-profile of TMC207 and moxifloxacin over time in the blood stream) will be evaluated by multiple blood samples from Day -1 tol Day 3. Participants in Group 1 will take a single 800-mg dose of TMC207 on Day 1 and a single dose of moxifloxacin placebo on Day 2 (Treatment A). Participants in Groups 2 and 3 will take a single dose of TMC207 placebo on Day 1 and a single 400-mg dose of moxifloxacin on Day 2 (Treatment B).¿ The study duration will be 3 days without screening and follow-up period included.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram, and clinical laboratory tests at screening
* A Body Mass Index of 18.0 to 28.0 kg/m2, extremes included
* Women must be postmenopausal for at least two years, be surgically sterile and must have negative serum pregnancy test at screening
* Non-smoking for at least three months prior to selection.

Exclusion Criteria:

* Infection with Hepatitis A, B, or C virus
* Infection with the human immunodeficiency virus (HIV)
* History of, or any current medical condition which could impact the safety of the participant in the study
* Previously participated in a TMC207 trial or received an investigational drug or vaccine within 60 days before the planned start of treatment
* A positive urine drug test at screening
* Volunteers with a clinically significant ECG abnormality or any other cardiac history (unusual T wave morphology, history of additional risk for Torsade de Pointes, electrolyte abnormalities, blood pressure outside of the normal range, or history of a clinically relevant heart rhythm disturbance or with a family history of Long QT Syndrome)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-02; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
ECG evaluation as a measure of QT and QTc interval | Measured Day -1 to Day 3

SECONDARY OUTCOMES:
ECG evaluation as a measure of non-QT interval electrocardiogram parameters (RR interval, HR, PR and QRS interval) | Measured on Day -1 until Day 3
Plasma concentrations of TMC207 and its N-monodesmethyl metabolite (M2) | Measured on Day -1 until Day 3
Evaluation of the concentration-effect relationship for QT/QTc for TMC207 and M2 | Measured on Day -1 until Day 3
Evaluation of the number of volunteers with adverse events, blood and urine tests, blood pressure and pulse tests, and ECGs as measures of safety and tolerability | Measured on Day -1 until Day 3 and Day 8-10 and 30 to 32 days after last study drug intake as safety follow up

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA